CLINICAL TRIAL: NCT04439487
Title: Thyromental Height Test as a New Method for Prediction of Difficult Intubation in Obese Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Piotr Palaczyński, Principal Investigator, Medical University of Silesia
Other Study IDs: TMHT-02
Record Dates: First submitted 2020-06-04; First posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Intubation, Intratracheal; Obesity; Predictive Value of Tests
Keywords: Difficult Intubation; Obesity; Thyromental Height Test
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obese patients requiring general anesthesia: Group consists of consecutive, adult, obese patients undergoing elective surgical procedures requiring general anaesthesia, direct laryngoscopy and intubation. All patients undergo general anesthesia according to a standardised protocol. They are preoxygenated with 100% oxygen breathed through a face mask for 3-5 minutes. Induction of general anaesthesia is achieved with propofol 1,5-2 mg·kg-1 (of Ideal Body Weight) and 0,1mg fentanyl or sufentanil 10µg. Muscle relaxation is accomplished with rocuronium 0.6 mg ·kg-1 (of Ideal Body Weight). Depth of muscular blockade is monitored using Train of Four (TOF) method. The first laryngoscopy attempt is performed at TOF 0. The patient is placed in an optimal, sniffing or ramped position as appropriate and a #3 or #4 Macintosh blade is used. Successful intubation is confirmed with bilateral auscultation and capnography.
  Interventions: Diagnostic Test: Anthropometric measurements during routine preoperative visit; Other: Assesment of intubation parameters during induction of general anaesthesia

INTERVENTIONS:
Diagnostic Test: Anthropometric measurements during routine preoperative visit — During routine preoperative anaesthetic visit and physical examination the following predictive test measurements are obtained by a research team member not involved in the further assessment of laryngoscopy: score in modified Mallampati test, Thyromental height, Sternomental distance, Thyromental distance, Neck circumference, Mouth opening distance
Other: Assesment of intubation parameters during induction of general anaesthesia — During induction of general anaesthesia and intubation research team member not involved in obtaining anthropometric measurements notes Number of intubation attempts, Intubation time, Subjective intubation difficulty, Use of bougie and Need of technique modification.

SUMMARY:
The main objective of this trial is to assess the clinical usefulness of thyromental height test (TMHT) in prediction of difficult intubation in obese patients scheduled for elective surgical procedures. The secondary aim is to evaluate usefulness of other commonly used predictive tests associated with difficult intubation in obese patients.

DETAILED DESCRIPTION:
Successful and fast intubation are crucial for the safety of general anaesthesia. Failed intubation and acute hypoxia remain among the major contributing factors of anaesthesia related deaths. Difficult intubation prevalence in literature is very inconsistent and varies between 1.5-20% of cases in general population, to even 50% in obese Thai population.

Obesity remains a challenging problem in perioperative care. It is assumed that the airway access may be restricted due to anatomic changes resulting from excess body weight. There are factors like diagnosed obstructive sleep apnoea or large neck circumference that also relate to occurrence of difficult intubation in obese patients.

There is a number of anthropometric scales and tests used for predicting difficult intubation in obese patients. However, none of them appears to be sensitive and specific enough to effectively predict difficult intubation.

Recently, simple and non-invasive test predicting difficult intubation was introduced-thyromental height test (TMHT). It shows promise as a more effective substitution for frequently cited anthropometric measures. It is based on the height between the anterior border of the thyroid cartilage and the anterior border of the mentum, measured while the patient lies in the supine position with closed mouth.

The main objective of this trial is to assess the clinical usefulness of TMHT in prediction of difficult intubation in obese patients scheduled for elective surgical procedures. The secondary aim is to evaluate usefulness of other commonly used predictive tests associated with difficult intubation in obese patients.

ELIGIBILITY:
Inclusion Criteria:

* qualification for elective surgical procedures, requiring general anaesthesia, direct laryngoscopy and intubation
* consent for participation in the trail
* age ≥18 years
* BMI ≥30 kg/m2

Exclusion Criteria:

* BMI ≤30 kg/m2
* patients overweight due to ascites or tumor
* emergency procedures
* visible anatomic abnormalities
* patients scheduled for awake fibreoptic intubation
* intubation failure
* lack of consent for participation in the trail

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Studied population will consist of consecutive obese, adult patients (BMI ≥30 kg/m2) qualified for elective surgical procedures, requiring general anaesthesia, direct laryngoscopy and intubation.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Score in Cormack-Lehane scale (CL). | Intraoperatively (an average of 5 minutes)
  During direct laryngoscopy after the induction of general anesthesia the laryngeal view is graded in Cormack-Lehane Scale by the laryngoscopist. Grade I is assigned when the glottis is fully visible, grade II when the glottis is partially visible, grade III when only the epiglottis is visible and grade IV when neither glottis nor epiglottis is visible.
Thyromental height (TMH). [mm] | Preoperatively (an average of 24 hours)
  Thyromental height is defined as the height between the anterior border of the thyroid cartilage (on the thyroid notch just between the 2 thyroid laminae) and the anterior border of the mentum (on the mental protuberance of the mandible). It is measured with a depth gauge during routine preoperative anaesthetic visit in supine position and closed mouth.

SECONDARY OUTCOMES:
Thyromental distance (TMD). [cm] | Preoperatively (an average of 24 hours)
  Thyromental distance is measured during routine preoperative visit as a height between the anterior border of the thyroid cartilage (on the thyroid notch just between the 2 thyroid laminae) and the anterior border of the mentum (on the mental protuberance of the mandible) with a depth gauge (21460605, Limit, Alingsås, Sweden) in millimetres, with the patient in supine position and closed mouth.
Sternomental distance (SMD). [cm] | Preoperatively (an average of 24 hours)
  Sternomental distance is measured during routine preoperative visit between the superior border of the manubrium sterni and the most anterior part of the mental prominence of the mandible with a tape measure (Standard, Hoechstmas, Sulzbach, Germany) as a distance in centimetres, with the patient in supine position, head fully extended, mouth closed.
Score in modified Mallampati test (MMT). | Preoperatively (an average of 24 hours)
  The oropharyngeal view is assessed according to modified Mallampati scale in sitting position, mouth maximally opened, tongue protruded, without phonation during routine preoperative anaesthetic visit. Grade I is assigned when the soft palate, uvula, fauces and pillars are fully visible, grade II when the soft palate, major part of uvula and fauces are visible, grade III when soft palate and base of uvula are visible and grade IV when only hard palate is visible.
Mouth opening (MO). [cm] | Preoperatively (an average of 24 hours)
  Mouth opening is measured as a distance between the lower and upper incisors with a tape measure (Standard, Hoechstmas, Sulzbach, Germany) in centimetres. Patients are in sitting position with mouth maximally opened, tongue retracted and without phonation.
Neck circumference (NC). [cm] | Preoperatively (an average of 24 hours)
  Neck circumference is measured at the level of the cricoid cartilage horizontally with a tape measure (Standard, Hoechstmas, Sulzbach, Germany) as a circumference in centimetres in the sitting position during routine preoperative visit.
Intubation time. [s] | Intraoperatively (an average of 5 minutes)
  Intubation time is defined as a time from direct laryngoscopy commencement to confirmation of endotracheal tube placement and noted during induction of general anaesthesia.
Intubation difficulty. | Intraoperatively (an average of 5 minutes)
  Subjective evaluation of intubation difficulty is noted during induction of general anaesthesia. Grade I is defined as an easy intubation, grade II a moderate intubation and grade III as a difficult intubation.
Number of intubation attempts. | Intraoperatively (an average of 5 minutes)
  Number of intubation attempts defined as a failed direct laryngoscopy without the use of endotracheal tube or insertion of endotracheal tube beyond the teeth line is noted during induction of general anaesthesia.
Use of bougie. | Intraoperatively (an average of 5 minutes)
  Necessity to use bougie during induction of general anaesthesia is noted.
Technique modification. | Intraoperatively (an average of 5 minutes)
  Necessity to modify technique of laryngoscopy or intubation is noted.

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - Medical University of Gdansk, Gdansk, Pomeranian Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny nr 1, Zabrze, Silesian Voivodeship